CLINICAL TRIAL: NCT03171961
Title: Effectiveness of Online Visit Compared With In-person Clinic Visit on Weight Loss in Overweight and Obese Women, a Randomized Clinical Trial
Brief Title: Effectiveness of Online Visit Compared With In-person Clinic Visit on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-207
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
Keywords: weight loss; Diet; online visit; clinic visit
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- online visit group (Experimental): in online visit group , subjects has online visit with dietitian every 2 weeks
  Interventions: Behavioral: online visit group
- clinic visit group (Experimental): clinic visit group ,subject has every 2 weeks in person visit at clinic
  Interventions: Behavioral: Clinic visit group
- self-directed group (Experimental): self-directed group ,subjects receive nutritional information via web and their energy needs for weight loss
  Interventions: Behavioral: self-directed group

INTERVENTIONS:
Behavioral: online visit group — subjects has online visit with dietitian every 2 weeks+diet
  Other Names: OV
  Arms: online visit group
Behavioral: Clinic visit group — Clinic visit group ,subjects has every 2 weeks in person visit at clinic+diet
  Other Names: CV
  Arms: clinic visit group
Behavioral: self-directed group — self-directed group receives nutritional information via web and their energy needs for weight loss
  Other Names: SD
  Arms: self-directed group

SUMMARY:
Online visit and online counseling via telemedicine technology is a new service for obese people who wish to lose weight but because of their active lifestyle and time limitation cannot come to clinic. The purpose of this study was to examine the efficacy this technology-based intervention on weight loss in obese and overweight female adults.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must be 18-45 years of age.
* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.
* Have access to the internet via broad- band ADSL or Mobile 4G

Exclusion Criteria:

* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medications that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
weight | 24 Weeks
  kg

SECONDARY OUTCOMES:
Waist circumference | 24 Weeks
  cm
Fasting blood glucose | 24 Weeks
  mmol/l
Fasting insulin level | 24 Weeks
  mU/l
HbA1c | 24 Weeks
  score
HOMA-IR | 24 Weeks
  Percentage (%)
lipid profiles | 24 Weeks
  mmol/l
liver function tests | 24 Weeks
  U/l

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - NovinDiet Clinic, Tehran
  - NovinDiet Clinic, Tehrān

IPD SHARING:
Plan to Share IPD: Undecided